CLINICAL TRIAL: NCT07081165
Title: Epidemiology of Tibial Plateau Fractures in a Tertiary Care Center: A Retrospective Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: National Trauma Center (Other)
Responsible Party: Principal Investigator, Sudeep Khanal, Doctor, National Trauma Center
Other Study IDs: TIBPLAT-NTC60
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-06

CONDITIONS: Tibial Plateau Fracture; Tibial Plateau Fractures
Keywords: Epidemiology; Fracture; Schatzker; Tibial Plateau; Trauma Center
MeSH Terms: conditions — Tibial Plateau Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective cross-sectional study was conducted following approval from the institutional review board. Patients who presented to our center over a four-year period, from July 1 2015 to June 30 2019, were included in the study. Participants were selected based on the inclusion and exclusion criteria following review of the medical records. A standardized proforma was used to collect the data and stored in Microsoft Excel. Data processing and analysis was done in Statistical Packages for the Social Sciences (SPSS) version 23.0. All categorical data were presented as percentages along with absolute numbers, while all continuous numerical data were reported as mean ± standard deviation. Tibial plateau fractures were classified according to Schatzker classification, which comprise six types, with severity increasing progressively from type I to type VI.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients presenting to hospital with diagnosis of tibial plateau fracture, regardless of age, sex, associated injuries and comorbidities. The diagnosis of tibial plateau fracture was confirmed after assessment of X-ray or Computed Tomography (CT) scan by an orthopedic surgeon.

Exclusion Criteria:

* The study excluded patients who presented with a tibia fracture other than a tibial plateau fracture, including proximal tibia fractures and isolated tibial spine fractures. Those with missing records (data or imaging) were excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included patients presenting to hospital with diagnosis of tibial plateau fracture, regardless of age, sex, associated injuries and comorbidities. The diagnosis of tibial plateau fracture was confirmed after assessment of X-ray or Computed Tomography (CT) scan by an orthopedic surgeon.
  The study excluded patients who presented with a tibia fracture other than a tibial plateau fracture, including proximal tibia fractures and isolated tibial spine fractures. Those with missing records (data or imaging) were excluded from the study.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Schatzker Classification | From July 2015 to June 2019

SECONDARY OUTCOMES:
Mode of Injury | From July 2015 to June 2019

IPD SHARING:
Plan to Share IPD: Undecided
IPD information can be shared if it is a reasonable request.